CLINICAL TRIAL: NCT07275437
Title: A Randomized, Controlled Trial Investigating the Effectiveness and Safety of Uptitration of Guideline Directed MEdical Therapy in Heart Failure With a Reduced Ejection Fraction With Limited Standardized Kidney Function Assessments (RESUME-HF-Kidney)
Brief Title: Effectiveness and Safety of Uptitration of Guideline Directed MEdical Therapy in Heart Failure With Reduced Ejection Fraction With Limited Kidney Function Assessments
Acronym: RESUME-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Onze Lieve Vrouwe Gasthuis (Other); Frisius Medisch Centrum (Other)
Responsible Party: Principal Investigator, Jozine ter Maaten, Assistant prof. J.M. ter Maaten, MD, PhD, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22833
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure; Heart Failure and Reduced Ejection Fraction; Heart Failure and Mildly Reduced Ejection Fraction
Keywords: Guideline-Directed Medical Therapy; Limited Kidney Function Assessments
MeSH Terms: conditions — Heart Failure; Heart Failure, Systolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Limited number of kidney function assessments (Experimental): Participants in this arm will have standardized kidney function assessments at baseline, three months, and six months. Kidney function assessments in between these moments will be blinded in the electronic patient dossier. Unblinding will be performed if the results are significantly abnormal.
  Interventions: Other: Blinded kidney function assessments
- Control (No Intervention): Participants will receive standard care, which includes frequent kidney function assessments.

INTERVENTIONS:
Other: Blinded kidney function assessments — Kidney function results will be blinded in the intervention group, except at baseline, three months, and six months.
  Arms: Limited number of kidney function assessments

SUMMARY:
Guideline-directed medical therapy (GDMT) for heart failure with reduced ejection fraction (HFrEF) constitutes of four medications that substantially reduce morbidity and mortality, and improve quality of life. In routine clinical practice, various physician- and patient-related factors lead to suboptimal initiation and uptitration of GDMT to optimal dosing, which is associated with worse patient outcomes. A perceived major barrier to the optimalization of GDMT are changes in kidney function and electrolytes, which prompts physicians to halt uptitration, reduce doses, or even discontinue GDMT. Changes in kidney function and electrolytes during optimalization of GDMT are common, but not associated with adverse events.

The hypothesis of this study is that a reduction in the number of kidney function assessments during initiation and uptitration of GDMT in HFrEF patients will lead to higher achieved doses of GDMT without safety concerns.

DETAILED DESCRIPTION:
Objective: To assess the effect of a reduction in kidney function assessments during optimalization of GDMT in patients with HFrEF on the achieved GDMT doses, safety, and clinical outcomes.

Study design: Randomized, controlled open-label study

Study population: 344 patients with new-onset or sub-optimally treated HFrEF referred to the outpatient clinic for optimalization of GDMT

Intervention (if applicable): Randomization to limited number of kidney function assessments or standard of care

Primary endpoint: The achieved average percentage dose of reno-active GDMT at 6 months relative to optimal dose.

Secondary endpoints: The achieved percentage dose of the individual reno-active GDMT drug classes at 6 months relative to optimal dose, and time to first occurrence of unplanned heart failure visit, heart failure hospitalization, or all-cause mortality till 9 months.

Safety endpoints: Incidence of doubling of creatinine, estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2, potassium >6 mmol/L, or potassium <3.5 mmol/L at any timepoint. An additional composite kidney endpoint is defined as a combination of hospitalization for kidney failure, dialysis or end-stage kidney disease (eGFR <15 mL/min/1.73 m2).

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to give written informed consent
2. Age ≥ 18 years
3. Diagnosed with HFrEF (LVEF≤ 45%) according to criteria from 2021 European Society of Cardiology guidelines for heart failure
4. Less than 100% target dose of 2 individual reno-active GDMT classes (ACEi/ARB/ARNI, MRA or SGLT-2i)

Exclusion Criteria:

1. eGFR<25 mL/min/1.73 m2 measured up to 30 days before the first visit
2. Potassium > 5.5 mmol/L or <3.5 mmol/L at screening
3. Known intolerance or allergy to two individual GDMT
4. Signs of hemodynamic instability and/or cardiogenic shock
5. Decompensated heart failure requiring treatment with intravenous loop diuretics
6. Known concomitant structural kidney disease such as polycystic kidney disease or renal artery stenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
The achieved average percentage dose of reno-active GDMT at 6 months relative to optimal dose. | 6 months

SECONDARY OUTCOMES:
The achieved percentage dose of the individual reno-active GDMT drug classes at 6 months relative to optimal dose. | 6 months
The time to first occurrence of unplanned heart failure visit, heart failure hospitalization, or all-cause mortality till 9 months. | 9 months

OTHER OUTCOMES:
The achieved average percentage dose of all GDMT at 6 months relative to optimal dose. | 6 months
Percentage change in NT-pro BNP at 6 months | 6 months
Percentage change in loop diuretics at 6 months | 6 months
Safety endpoint | Till 6 months
  Incidence of doubling of creatinine, estimated glomerular filtration rate (eGFR) <20 mL/min/1.73 m2, potassium >6 mmol/L, or potassium <3.5 mmol/L
Composite kidney endpoint | 6 months
  Hospitalization for kidney failure, dialysis or end-stage kidney disease (eGFR <15 mL/min/1.73 m2).

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Onze Lieve Vrouwe Gasthuis, Amsterdam, North Holland
  - Frisius MC, Leeuwarden, Provincie Friesland

IPD SHARING:
Plan to Share IPD: Undecided